CLINICAL TRIAL: NCT06482021
Title: Comparative Effectiveness Of Low Extra-Corporeal Shock Wave Versus Acetylcholine Iontophoresis On Type2 Diabetic Neuropathy: Randomized Clinical Trial
Brief Title: Comparative Effectiveness Of Low Extra-Corporeal Shock Wave Versus Acetylcholine Iontophoresis On Type2 Diabetic Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ibrahim Abuzaid, Director, Head of Department of Physiotherapy for Cardiovascular/Respiratory and Geriatrics, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Comparative Study
Record Dates: First submitted 2024-06-08; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Nephropathy
Keywords: Acetylcholine iontophoresis, shockwave
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Intervention Model Description: the study will be designed to compare the effect of extracorporeal shock wave therapy and acetylcholine iontophoresis on microcirculation changes as a possible new therapy for type 2 diabetic peripheral neuropathy.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (A) Low-intensity shock wave group (Experimental): Study group A will receive low-intensity extracorporeal shock wave therapy Li-ESWT (3 Hz, 0.09 mJ/mm2, 300 pulses), for two sessions per week for six weeks. Nitric oxide level and the electrophysiology (EMG) of peripheral nerves and muscles were measured pre and post-treatment.
  Interventions: Device: Low-intensity extracorporeal shock wave
- Study group (B) Acetylcholine iontophoresis group (Experimental): Study group (B) will receive iontophoresis by acetylcholine current intensity of 3 to 5 mA. Check skin every 3-5 minutes for signs of skin irritation with (15) min for three sessions per week for six weeks. Nitric oxide level and the electrophysiology (EMG) of peripheral nerves and muscles were measured pre and post-treatment.
  Interventions: Device: Low-intensity extracorporeal shock wave

INTERVENTIONS:
Device: Low-intensity extracorporeal shock wave — Acetylcholine iontophoresis• The Iontophoresis comprises of electric impulses from a low voltage galvanic current stimulation unit to drive ions (Ach) (1%) into soft tissue structures.
  Other Names: Device, ASTAR Swit 33, 43-382 dual-channel Stimulator (Bielsko-Biata, Poland) 230V-, 50/60 HZ, max 70 W, 100VA, was used.

SUMMARY:
In our thesis, we will compare the effectiveness of low-intensity shock wave versus acetylcholine iontophoresis as a possible new therapy for microcirculation changes in type 2 diabetic neuropathy

DETAILED DESCRIPTION:
Methods: A group of 80 patients (male and female) diagnosed with type 2 diabetes mellitus, was included in the study. Their age ranged from 40-60 years. Patients randomly will be divided into two groups: Study groups (A) 40 patients with type 2 diabetes mellitus with clinically proven peripheral neuropathy. And study group (B) 40 patients with type 2 diabetes mellitus with clinically proven peripheral neuropathy. They were selected from South Valley University Hospitals. Group A received low-intensity extracorporeal shock wave therapy Li-ESWT (3 Hz, 0.09 mJ/mm2, 300 pulses), for two sessions per week for six weeks. Study group (B) received iontophoresis by acetylcholine current intensity of 3 to 5 mA. Check skin every 3-5 minutes for signs of skin irritation with (15) min for three sessions per week for four weeks. Nitric oxide level and the electrophysiology (EMG) of peripheral nerves and muscles were measured pre and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients have to be symptomatically stable with type 2 diabetes mellitus complicated with peripheral neuropathy.
* Optimized pharmacological treatment that will be remained unchanged throughout the study.

Exclusion Criteria:

* Implanted cardiac pacemakers.
* Patients with known skin allergies.
* Presence of skin inflammations.
* Peripheral vascular disease.
* Patients with unstable angina pectoris.
* Progressive ventricular dysrhythmia.
* Intermittent claudication.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological investigations of peripheral nerves (latency, amplitude and velocity of peripheral nerves) | Six weeks
  Electrophysiological investigations of peripheral nerves were measured pre and post treatment for both groups (latency, amplitude and velocity of peripheral nerves)

SECONDARY OUTCOMES:
Nitric oxide laboratories for measurement of nitric oxide level | Six weeks
  Nitric oxide laboratories for measurement of nitric oxide level were measured pre and post treatment for both groups.

IPD SHARING:
Plan to Share IPD: Undecided
After publication

REFERENCES:
- [Result] Chen KT, Chen YP, Kuo YJ, Chiang MH. Extracorporeal Shock Wave Therapy Provides Limited Therapeutic Effects on Carpal Tunnel Syndrome: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2022 May 19;58(5):677. doi: 10.3390/medicina58050677. PMID 35630095
- [Result] Melese H, Alamer A, Getie K, Nigussie F, Ayhualem S. Extracorporeal shock wave therapy on pain and foot functions in subjects with chronic plantar fasciitis: systematic review of randomized controlled trials. Disabil Rehabil. 2022 Sep;44(18):5007-5014. doi: 10.1080/09638288.2021.1928775. Epub 2021 May 26. PMID 34038642